CLINICAL TRIAL: NCT05659160
Title: Triage of Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions-2 (TRACK-LVO-2): an Imaging-based Patient Registry Study
Brief Title: Triage of Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions-2
Acronym: TRACK-LVO-2
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2022-WM12
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute Ischemic; Endovascular Procedures; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke; Endovascular Therapy; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular therapy: Timely thrombectomy for acute ischemic stroke patients with large vessel occlusion by either stent retriever, thrombus aspiration, others, or combination methods.
  Interventions: Procedure: Endovascular Therapy
- Best medical management: Patients enrolled in this group received the best medical management.

INTERVENTIONS:
Procedure: Endovascular Therapy — Endovascular therapy, as an adjunct to standard stroke therapy, may be beneficial for a very select population of patients who present with an acute ischemic stroke and have a proven large, proximal occlusion on imaging.
  Endovascular therapy includes any one or more of the following:
  Intra-arterial thrombolytic therapy, aspiration, stent retrieval, or a combination of multiple mechanical devices.
  Groups: Endovascular therapy

SUMMARY:
The objective of this study is to create a comprehensive, real-world, multi-center observational registry of consecutive patients admitted to hospitals with acute ischemic stroke (AIS) caused by large vessel occlusions (LVO), who are treated with either endovascular therapy (EVT) or the best available medical management (BMM).

DETAILED DESCRIPTION:
The TRACK-LVO registry is an observational study conducted across multiple centers with the aim of improving the detection and treatment of large vessel occlusion (LVO) in acute ischemic stroke (AIS) patients. LVO is a major predictor of unfavorable outcomes in stroke patients, and the most effective imaging modalities for its detection remain a topic of debate.

To address this, the investigators will enroll consecutive AIS patients with LVO screened under different imaging modalities and compared the efficacy of endovascular therapy (EVT) and best medical management (BMM). The registry defines LVO as an occlusion of the intracranial ICA with or without the involvement of the terminal bifurcation, M1 and/or M2 segment of the MCA, A1 and/or A2 segment of the ACA, VA, BA, or P1 and/or P2 segment of the PCA. Patient information, including basic demographic profiles, imaging characteristics such as volume of ischemic core and occlusion site, and treatment-related complications will be collected for both EVT and BMM groups. For patients in the EVT group, detailed information on the EVT procedure and angiographic images will also be collected.

The study aims to identify the optimal imaging modalities for LVO detection and to compare the prognosis of AIS patients with LVO receiving EVT versus BMM. This academic, real-world, multi-center, observational registry will contribute valuable insights to improve the detection and treatment of LVO in AIS patients, ultimately improving patient outcomes and reducing the burden of stroke on public health and socio-economic development.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted from Jan. 1st 2018 to Jan. 1st 2028;
2. Age ≥ 18;
3. Ischemic stroke confirmed by head CT or MRI;
4. Large vessel occlusion confirmed by head CTA or MRA: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA), and posterior cerebral artery (PCA P1/P2);
5. Patients receiving either endovascular therapy or best medical treatment;

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute ischemic stroke patients with large vessel occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified ranking scale (mRS) at 90 days | 90 days
  A 0-6 scale running from perfect health without symptoms to death.
Mortality within 90 days | 90 days
  mortality of any causes.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) scores at 90 days | 90 days
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Occurrence of periprocedural complications | 14 days postoperatively
  Periprocedural complications include any intracranial hemorrhage, cerebral edema, brain herniation and pneumonia.
ASPECT (Alberta Stroke Program Early CT score) | Day 0
  ASPECTS is a 10-point quantitative topographic CT scan score used in patients with middle cerebral artery (MCA) stroke.
EuroQol five dimensions questionnaire (EQ-5D) | 1 year
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Sencond Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Beijing University Binhai Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided